CLINICAL TRIAL: NCT07308938
Title: Trial of Topical Fluorometholone as Adjunctive Therapy for Bacterial Corneal Ulcers
Brief Title: Fluorometholone Study
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vishal Jhanji (Other)
Collaborators: University of Pittsburgh Medical Center (Other)
Responsible Party: Sponsor-Investigator, Vishal Jhanji, Professor of Ophthalmology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY25110161
Record Dates: First submitted 2025-12-26; First posted 2025-12-30 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Keratitis Bacterial; Corneal Ulcer (Diagnosis)
MeSH Terms: conditions — Corneal Ulcer; Disease | interventions — Fluorometholone

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, parallel-group clinical cohort study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Experimental): Standard Topical Antibiotic Therapy + Fluorometholone
  Interventions: Drug: Adjunctive Topical Fluorometholone (FML) 0.1%; Drug: Standard Topical Antibiotic Therapy
- Control Arm (Active Comparator): Standard Topical Antibiotic Therapy Alone
  Interventions: Drug: Standard Topical Antibiotic Therapy

INTERVENTIONS:
Drug: Adjunctive Topical Fluorometholone (FML) 0.1% — Adjunctive Topical Fluorometholone (FML) 0.1% will be used
  Arms: Intervention Arm
Drug: Standard Topical Antibiotic Therapy — Patients will be treated with antibiotics (Cefazolin, Tobramycin or Moxifloxacin) we per treating physician

SUMMARY:
The investigators seek to determine whether adjunctive topical fluorometholone (FML) improves best-corrected visual acuity (BCVA) at 3 months in patients with bacterial corneal ulcers compared with standard topical antibiotic therapy alone.

DETAILED DESCRIPTION:
In this prospective, randomized, parallel-group clinical cohort study, the investigators seek to determine whether adjunctive topical fluorometholone (FML) improves best-corrected visual acuity (BCVA) at 3 months in patients with bacterial corneal ulcers compared with standard topical antibiotic therapy alone. The primary objective is to compare the mean 3-month BCVA (logMAR) between the intervention arm (standard topical antibiotic therapy + FML 0.1%) and a control arm (standard topical antibiotic therapy alone).

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged ≥ 18 years.
2. Clinical diagnosis of a bacterial corneal ulcer based on slit-lamp examination.
3. Ulcer severity classified as:

   * Mild: Diameter ≤ 3 mm AND stromal depth ≤ 1/3 thickness.
   * Moderate: Diameter >3-6 mm and/or stromal depth > 1/3-2/3.
   * Severe: Diameter >6 mm and/or stromal depth >2/3.
4. Completed microbiologic work-up including ≥ 1 of:

   * Corneal culture, or
   * PCR testing.
5. Received ≥ 48-96 hours of empiric topical antibiotic therapy prior to randomization (fluoroquinolone monotherapy or fortified cefazolin/tobramycin based on standard of care).
6. Able and willing to provide informed consent and comply with study visits.

Exclusion Criteria:

1. Clinical or laboratory evidence of:

   * Herpes simplex keratitis.
   * Acanthamoeba keratitis.
   * Fungal keratitis (positive smear, culture or PCR).
2. Corneal perforation or imminent perforation at presentation.
3. Current use of:

   * Topical corticosteroids in the study eye, or
   * Systemic corticosteroids during this ulcer episode.
4. History of steroid-responsive glaucoma or uncontrolled intraocular pressure (IOP).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity (BCVA) | From enrollment to 3 months
  BCVA (logMAR) at 3 months post-randomization in the study eye.

SECONDARY OUTCOMES:
Visual Improvement | From enrollment (Day 1) to Week 1, Month 1, Month 3.
  Change in BCVA from baseline to weeks 1 and 4, and 3 months.
Time to re-epithelialization | From enrollment to 3 months
  Time to re-epithelialization
Intraocular Pressure (IOP) | From enrollment (Day 1) to Day 3, 1 Week, 1 Month, 3 Months.
  IOP measurements at all follow-up visits.
Complications | From enrollment to Month 3.
  Progressive thinning or perforation; hypopyon development or increase; endophthalmitis; fibrin formation; or worsening infiltrate size or depth ≥50%.

CONTACTS AND LOCATIONS:
Overall Officials: Vishal Jhanji, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Vision Institute, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
The data would be made available upon reasonable request.